CLINICAL TRIAL: NCT06057012
Title: A Phase 2a, Multicenter, Open-label Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Descriptive Efficacy of BRII-296 in Adults With Severe Postpartum Depression (PPD)
Brief Title: A Study of BRII-296 in Adults With Severe Postpartum Depression (PPD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Brii Biosciences Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BRII-296-002
Record Dates: First submitted 2023-09-21; First posted 2023-09-28 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Severe Postpartum Depression
Keywords: Treatment
MeSH Terms: conditions — Depression, Postpartum | interventions — Methylprednisolone Acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- BRII-296 + Depo Medrol (Experimental): Participants will receive BRII-296 600 milligram (mg) and Depo Medrol (80 milligram per milliliter [mg/mL]) on Day 1 as a combination therapy.
  Interventions: Drug: BRII-296; Drug: Depo Medrol

INTERVENTIONS:
Drug: BRII-296 — BRII-296 will be given via intramuscular injection.
Drug: Depo Medrol — Depo Medrol will be given via intramuscular injection.

SUMMARY:
The primary purpose of this study is to evaluate the safety and tolerability of BRII-296 administered by 2 intramuscular injections, administered with Depo Medrol as assessed by the incidence of adverse events, changes from baseline in vital signs, pulse oximetry, clinical laboratory evaluations, electrocardiograms (ECGs), Stanford Sleepiness Scale (SSS), Glasgow Coma Scale (GCS) in conjunction with clinical assessment, and suicidal ideation using the Columbia Suicide Severity Rating Scale (C-SSRS).

ELIGIBILITY:
Inclusion Criteria:

* Participant either must have ceased lactating at screening or is still lactating actively breastfeeding at screening , must agree temporarily cease giving breast milk to her infant(s)
* Participant has had a Major Depressive Episode that began no earlier than the third trimester and no later than the first 4 weeks following delivery, as diagnosed by the Structured Clinical Interview for Diagnostic and Statistical Manual of Mental Disorders (DSM-5)
* Participant was <12 months postpartum
* Participant is amenable to intramuscular administration of investigational product on Day 1 and remaining inpatient until at least Day 4

Exclusion Criteria:

* Active psychosis
* Attempted suicide associated with current episode of postpartum depression
* Medical history of seizures
* Medical history of bipolar disorder, schizophrenia, and/or schizoaffective disorder

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2023-09-29 (Actual); Primary Completion 2024-03-13 (Actual); Study Completion 2024-03-13 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs) | From the first dose of study drug up to Day 45
Number of Participants With Adverse Events (AEs) According to Severity | From the first dose of study drug up to Day 45
  Severity will be assessed according to the following scale: Mild, moderate and severe.
Number of Participants With Change From Baseline in Clinically Significant Vital Sign Parameters | Baseline up to Day 45
Number of Participants With Abnormal Electrocardiogram (ECG) Parameters | From the first dose of study drug up to Day 45
Number of Participants With Change From Baseline in Clinically Significant Clinical Laboratory Evaluations | From the first dose of study drug up to Day 45
Number of Participants With Columbia-Suicide Severity Rating Scale (C-SSRS) Responses | Baseline up to Day 45
  The suicidal ideation and behavior will be monitored during the study using the C-SSRS. This scale consists of a "Baseline/Screening" version that assesses the lifetime and recent experience of the participant with suicidal ideation and behavior, and a "Since Last Visit" version that focuses on suicidality since the last study visit. The C-SSRS includes "yes" or "no" responses for assessment of suicidal ideation and behavior as well as numeric ratings for severity of ideation, if present (from 1 to 5, with 5 being the most severe).
Change From Baseline in Glasgow Coma Scale (GCS) Score | Baseline up to Day 45
  The GCS is a simple measure of the depth and duration of impaired consciousness and coma. 3 domains of alertness will be evaluated: eye opening response (scored 1 [None] to 4 [Spontaneous]), verbal response (scored 1 [None] to 5 [Oriented]), and motor response (scored 1 [None] to 6 [Obeys commands]). Total scores range from 3 to 15, with 15 reflecting full alertness.
Change From Baseline in Stanford Sleepiness Scale (SSS) Score | Baseline up to Day 45
  The SSS is a participant-rated measure of sleepiness, frequently used for both research and clinical purposes. The SSS evaluates sleepiness at specific moments in time. Respondents rate their current degree of sleepiness and alertness on a scale of 1 to 7, where the lowest score of '1' indicates the respondent is 'feeling active, vital, alert, or wide awake' and the highest score of '7' indicates the respondent is 'no longer fighting sleep, sleep onset soon; having dream-like thoughts'.
PK of Brexanolone: Maximum Observed Plasma Concentration (Cmax) | Day 1- Day 45
PK of Brexanolone: Time to Reach Cmax (Tmax) | Day 1- Day 45
PK of Brexanolone: Area Under the Concentration-time Curve From Time 0 to Last Measurable Concentration (AUC0-last) | Day 1- Day 45
PK of Brexanolone: Area Under the Concentration-time Curve From Time 0 to Infinity (AUC0-inf) | Day 1- Day 45
PK of Brexanolone: Apparent Terminal Elimination Half-life (t½) | Day 1- Day 45
PK of Brexanolone: Apparent Clearance (CL/F) | Day 1- Day 45
PK of Brexanolone: Volume of Distribution (Vz/F) | Day 1- Day 45

SECONDARY OUTCOMES:
Change From Baseline in Hamilton Depression Rating Scale (HAM-D) Total Score | Baseline and at Days 2, 3, 4, 8, 15, 30, and 45
  The 17-item HAM-D will be used to rate the severity of depression in participants who are already diagnosed as depressed. The 17-item HAM-D is comprised of individual ratings related to the following symptoms: depressed mood (sadness, hopeless, helpless, and worthless), feelings of guilt, suicide, insomnia (early, middle, and late), work and activities, retardation (slowness of thought and speech, impaired ability to concentrate, and decreased motor activity), agitation, anxiety (psychic and somatic), somatic symptoms (gastrointestinal and general), genital symptoms, hypochondriasis, loss of weight, and insight. The total scores range from 0-52. Higher score indicates more depression.
Number of Participants With HAM-D Response | Baseline and at Days 2, 3, 4, 8, 15, 30, and 45
  Response is defined as >=50 percent (%) reduction from baseline in HAM-D total score. The HAM-D is a 17-item scale used to rate the severity of depression in participants who are already diagnosed as depressed. The total scores of HAM-D range from 0-52. Higher score indicates more depression.
Number of Participants With HAM-D Remission | Baseline and at Days 2, 3, 4, 8, 15, 30, and 45
  Remission is defined as <=7.0 HAM-D total score. The HAM-D is a 17-item scale used to rate the severity of depression in participants who are already diagnosed as depressed. The total scores of HAM-D range from 0-52. Higher score indicates more depression.
Number of Participants With Clinical Global Impression - Improvement (CGI-I) Response | Baseline and at Days 2, 3, 4, 8, 15, 30, and 45
  The CGI-I item employs a 7-point Likert scale to measure the overall improvement in the participant's condition posttreatment. The clinician will rate the participant's total improvement, whether or not it is due entirely to investigational product treatment. Response choices include: 0 = not assessed, 1 = very much improved, 2 = much improved, 3 = minimally improved, 4 = no change, 5 = minimally worse, 6 = much worse, and 7 = very much worse. CGI-I response will be defined as having a CGI-I score of "very much improved" or "much improved."
Change From Baseline in Clinical Global Impression - Severity (CGI-S) Response | Baseline and at Days 2, 3, 4, 8, 15, 30, and 45
  The CGI-S item uses a 7- point Likert scale to rate the severity of the patient's illness at the time of assessment, relative to the clinician's past experience with patients who have the same diagnosis. Considering total clinical experience, a patient is assessed on severity of mental illness at the time of rating. Choices include: 1 = normal, not at all ill; 2 = borderline mentally ill; 3 = mildly ill; 4 = moderately ill; 5 = markedly ill; 6 = severely ill; and 7 = extremely ill.
Change From Baseline in HAM-D Bech-6 Subscale Score | Baseline and at Days 2, 3, 4, 8, 15, 30, and 45
  The HAM-D Bech 6 subscale score is calculated as the sum of the following six items: Item # 1 (depressed mood), Item # 2 (feelings of guilt), Item # 7 (work and activities), Item # 8 (retardation), Item # 10 (anxiety psychic), and Item # 13 (general somatic symptoms). Each item is scored in a range of 0 to 2 or 0 to 4, with higher scores indicating a greater degree of depression. The scores will be transformed to a 100-point scale with a higher score indicating a greater degree of depression. A negative change from baseline indicates less depression. A positive change from baseline indicates more depression.
Change From Baseline in HAM-D Individual Item Score | Baseline and at Days 2, 3, 4, 8, 15, 30, and 45
  The HAM-D comprises individual ratings of the following symptoms scored in a range of 0 to 2: insomnia (early, middle, late), somatic symptoms (gastrointestinal and general), genital symptoms, loss of weight, and insight. The following symptoms are scored in a range of 0 to 4: agitation, depressed mood, feelings of guilt, suicide, work and activities, retardation, anxiety (psychic and somatic), and hypochondriasis. Higher scores indicate a greater degree of depression. A negative change from baseline indicates less depression. A positive change from baseline indicates more depression.
Change From Baseline in Hamilton Anxiety Rating Scale (HAM-A) Total Score | Baseline and at Days 2, 3, 4, 8, 15, 30, and 45
  The 14-item HAM-A will be used to rate the severity of symptoms of anxiety. Each of the 14 items is defined by a series of symptoms and measures both psychic anxiety (mental agitation and psychological distress) and somatic anxiety (physical complaints related to anxiety). Scoring for the HAM-A is calculated by assigning scores of 0 (not present) to 4 (very severe), with a total score range of 0 to 56, where less than (<) 17 indicates mild severity, 18 to 24 mild to moderate severity, and 25 to 30 moderate to severe severity. The HAM-A total score will be calculated as the sum of the 14 individual item scores.

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - Cenexel CNR, Sherman Oaks, California
  - CenExel CNS-Torrance, Torrance, California
  - Clinical Research Center of Florida, Boynton Beach, Florida
  - Aventura Clinical Research, LLC, Davie, Florida
  - South Florida Research Phase I-IV Inc, Miami Springs, Florida
  - Synexus Clinical Research US, Inc., Atlanta, Georgia
  - Cenexel ACMR Atlanta Center for Medical Research, Atlanta, Georgia
  - iResearch Atlanta, LLC, Decatur, Georgia
  - Research Carolina Elite, Denver, North Carolina
  - North Texas Clinical Trials, Fort Worth, Texas
  - Maximos OB/GYN, League City, Texas

IPD SHARING:
Plan to Share IPD: Undecided